CLINICAL TRIAL: NCT03971916
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Doses of HBM9161(HL161BKN) in Healthy Chinese Volunteers (Randomized, Single-blinded, Placebo-controlled Trial)
Brief Title: A Phase I Study Evaluating the Safety, Tolerability, PK and PD in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Harbour BioMed (Guangzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: 9161.1
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Healthy Chinese Volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HBM9161 340mg (Experimental)
  Interventions: Drug: HBM9161(HL161BKN)
- HBM9161 510mg (Experimental)
  Interventions: Drug: HBM9161(HL161BKN)
- HBM9161 680mg (Experimental)
  Interventions: Drug: HBM9161(HL161BKN)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HBM9161(HL161BKN) — Subcutaneous injection; Single dose on Day 1
  Arms: HBM9161 340mg; HBM9161 510mg; HBM9161 680mg
Drug: Placebo — Subcutaneous injection; Single dose on Day 1
  Arms: Placebo

SUMMARY:
Trial Objective: To investigate the safety, tolerability, PK, and PD following single ascending doses of HBM9161 in healthy Chinese subjects.

DETAILED DESCRIPTION:
HBM9161(HL161BKN) is a human monoclonal antibody. HBM9161 targets the neonatal Fc receptor (FcRn) . The neonatal FcRn is a potential therapeutic target for many autoimmune diseases. This Phase I study will evaluate the safety, tolerability, PK, and PD of subcutaneous (SC) doses of HBM9161(HL161BKN) (abbreviated as HBM9161) in healthy Chinese subjects. Up to 24 healthy Chinese subjects will be randomized into the study. For each dose group, 8 subjects will be randomized (6 subjects to HBM9161 group and 2 subjects to placebo group).

This study will also provide guidance on doses to be used in future studies involving patients with autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Han Chinese male or female subjects, and his/her biological parents and grandparents are of Han Chinese ethnicity.
2. Body weight ≥ 50kg with BMI ≥19.0 and <=24.0 kg/m2 at screening and baseline visit.
3. Generally, in good health with no clinically significant abnormalities as determined by medical history, physical examination, 12-lead ECG and clinical laboratory tests.

Exclusion Criteria:

1. Subject has a total IgG level of < 700mg/dL at screening.
2. Subject has an active infection or has had a serious infection within 6 weeks prior to Day -1 or infection requiring oral anti-infective agents within 2 weeks prior to Day-1, or subject had a febrile illness or symptomatic, viral, bacterial, or fungal infection within 1 week prior to admission (Day -1).
3. History of relevant allergy/hypersensitivity (including allergy to study drug or its excipients).
4. Any laboratory values outside the reference range that are of clinical significance according to investigator's clinical judgement.
5. Subject has estimated creatinine clearance ≤ 80 mL/min calculated by Cockcroft Gault formula at screening.
6. Subject has any ECG abnormality defined in the protocol (a single repeat will be allowed for eligibility determination) at screening or Day -1:
7. Positive HIV test result at screening.
8. Positive testing for HBs Antigen and/or a positive Hepatitis C antibody test result at screening.
9. Subject has a positive T-cell interferon-γ release assay (TIGRA) result
10. Subjects who had immunization within 4 weeks before screening; or subjects who plan to have immunization during the study and within 12 weeks after dosing of the study drug.
11. For female subjects, positive pregnancy test at screening or Day -1, or planning to become pregnant from screening until 90 days after the dosing of the study drug.
12. Lactating female subjects.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-11-06 (Actual)

PRIMARY OUTCOMES:
The number [N (%)] of subjects with drug-related AEs | 85 days
  The number [N (%)] of subjects with drug-related AEs

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Yat Hin YAP, Principal Investigator — Queen Mary Hospital, Phase 1 Clinical Trials Centre
Locations (1):
- Queen Mary Hospital, Phase 1 Clinical Trials Centre, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No